CLINICAL TRIAL: NCT06119581
Title: SUNRAY-01, A Global Pivotal Study in Participants With KRAS G12C-Mutant, Locally Advanced or Metastatic Non-Small Cell Lung Cancer Comparing First-Line Treatment of LY3537982 and Pembrolizumab vs Placebo and Pembrolizumab in Those With PD-L1 Expression ≥50% or LY3537982 and Pembrolizumab, Pemetrexed, Platinum vs Placebo and Pembrolizumab, Pemetrexed, Platinum Regardless of PD-L1 Expression
Brief Title: A Study of First-Line Olomorasib (LY3537982) and Pembrolizumab With or Without Chemotherapy in Patients With Advanced KRAS G12C-Mutant Non-small Cell Lung Cancer
Acronym: SUNRAY-01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18612; J3M-MC-JZQB (Other: Eli Lilly and Company); U1111-1288-0565 (Other: Universal Trial Number); 2023-503412-33-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis
Keywords: Advanced Non-Small Cell Lung Cancer; KRAS G12 Lung Cancer; Advanced Lung Cancer; Metastatic Lung Cancer; KRAS G12C inhibitor; KRAS G12C Positive; KRAS Mutation; KRAS G12 Mutation; Lung Cancer Mutation; Olomorasib; Lung Diseases; Neoplastic Processes; Pathologic Processes; Neoplasm Metastasis; Non-Small Cell Lung Cancer; Non-Small Cell Lung Cancer (NSCLC); Antineoplastic Agents; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms; Lung Diseases; Neoplastic Processes; Pathologic Processes; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms | interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Optimization: LY3537982 Dose Level 1 plus Pembrolizumab (Experimental): LY3537982 Dose level 1 administered orally in combination with pembrolizumab administered intravenously (IV) in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: LY3537982; Drug: Pembrolizumab
- Dose Optimization: LY3537982 Dose Level 2 plus Pembrolizumab (Experimental): LY3537982 Dose level 2 administered orally in combination with pembrolizumab administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: LY3537982; Drug: Pembrolizumab
- Safety Lead In: LY3537982 plus Pembrolizumab, Pemetrexed and Platinum (Experimental): LY3537982 administered orally in combination with pembrolizumab, pemetrexed, and platinum (cisplatin or carboplatin) administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: LY3537982; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- Part A: LY3537982 plus Pembrolizumab (Experimental): LY3537982 administered orally in combination with pembrolizumab administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: LY3537982; Drug: Pembrolizumab
- Part A: Placebo plus Pembrolizumab (Placebo Comparator): Placebo administered orally in combination with pembrolizumab administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Pembrolizumab; Drug: Placebo
- Part B: LY3537982 plus Pembrolizumab, Pemetrexed, and Platinum (Experimental): LY3537982 administered orally in combination with pembrolizumab, pemetrexed, and platinum (cisplatin or carboplatin) administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: LY3537982; Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- Part B: Placebo plus Pembrolizumab, Pemetrexed, and Platinum (Placebo Comparator): Placebo administered orally in combination with pembrolizumab, pemetrexed, and platinum (cisplatin or carboplatin) administered IV in 21-day cycles. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Pembrolizumab; Drug: Placebo; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: LY3537982 — Administered orally.
  Other Names: Olomorasib
  Arms: Dose Optimization: LY3537982 Dose Level 1 plus Pembrolizumab; Dose Optimization: LY3537982 Dose Level 2 plus Pembrolizumab; Part A: LY3537982 plus Pembrolizumab; Part B: LY3537982 plus Pembrolizumab, Pemetrexed, and Platinum; Safety Lead In: LY3537982 plus Pembrolizumab, Pemetrexed and Platinum
Drug: Pembrolizumab — Administered IV.
Drug: Placebo — Administered orally.
  Arms: Part A: Placebo plus Pembrolizumab; Part B: Placebo plus Pembrolizumab, Pemetrexed, and Platinum
Drug: Cisplatin — Administered IV.
  Arms: Part B: LY3537982 plus Pembrolizumab, Pemetrexed, and Platinum; Part B: Placebo plus Pembrolizumab, Pemetrexed, and Platinum; Safety Lead In: LY3537982 plus Pembrolizumab, Pemetrexed and Platinum
Drug: Carboplatin — Administered IV.
  Arms: Part B: LY3537982 plus Pembrolizumab, Pemetrexed, and Platinum; Part B: Placebo plus Pembrolizumab, Pemetrexed, and Platinum; Safety Lead In: LY3537982 plus Pembrolizumab, Pemetrexed and Platinum
Drug: Pemetrexed — Administered IV.
  Arms: Part B: LY3537982 plus Pembrolizumab, Pemetrexed, and Platinum; Part B: Placebo plus Pembrolizumab, Pemetrexed, and Platinum; Safety Lead In: LY3537982 plus Pembrolizumab, Pemetrexed and Platinum

SUMMARY:
The purpose of this study is to assess if adding LY3537982 (olomorasib) in combination with standard of care anti-cancer drugs is more effective than standard of care in participants with untreated advanced NSCLC. NSCLC must have a change in a gene called KRAS G12C. Study participation, including follow-up, could last up to 3 years, depending on how you and your lung cancer are doing.

DETAILED DESCRIPTION:
Dose Optimization, Part A, and Part B are randomized. Safety Lead-In for Part B is single arm, non-randomized.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC with Stage IIIB-IIIC or Stage IV disease, not suitable for curative intent radical surgery or radiation therapy.
* Part B and Safety Lead-In Part B: the histology of the tumor must be predominantly non-squamous (in line with pemetrexed label).
* Must have disease with evidence of KRAS G12C mutation.
* Must have known programmed death-ligand 1 (PD-L1) expression

  * Part A: Greater than or equal to (≥)50 percent (%).
  * Part B: 0% to 100%.
* Must have measurable disease per RECIST v1.1.
* Must have an ECOG performance status of 0 or 1.
* Estimated life expectancy ≥12 weeks.
* Ability to swallow capsules.
* Must have adequate laboratory parameters.
* Contraceptive use should be consistent with local regulations for those participating in clinical studies.
* Women of childbearing potential must

  * Have a negative pregnancy test.
  * Not be breastfeeding during treatment

Exclusion Criteria:

* Have a documented additional validated targetable oncogenic driver mutation or alteration in genes such as epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), BRAF (V600E), human epidermal growth factor receptor 2 (HER2), MET (exon 14), ROS1, rearranged during transfection (RET), or neurotrophic tyrosine receptor kinase (NTRK)1/2/3.
* Have had any of the following prior to randomization:

  -- Prior systemic therapy (chemotherapy, immunotherapy, targeted therapy, or biological therapy) for advanced or metastatic NSCLC.

  --- 1 cycle of standard-of-care treatment prior to study enrollment will be allowed for cases where immediate treatment is clinically indicated:
* Have known active central nervous system metastases and/or carcinomatous meningitis.

Exclusion Criteria for Participants receiving Pemetrexed and Platinum (Part B and Safety Lead-In Part B)

* Have predominantly squamous cell histology for NSCLC
* Only for participants with mild to moderate renal insufficiency: Unable to avoid aspirin, ibuprofen, or other nonsteroidal anti-inflammatory drugs (NSAIDs) two days before (5 days for long acting NSAIDs), day of, and two days after administration of pemetrexed
* Is unable or unwilling to take folic acid or vitamin B12 supplementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1016 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Dose Optimization and Safety Lead-In Part B: Number of Participants with a Treatment Emergent Adverse Event(s) (TEAE) | Randomization to first documented progression of disease or death from any cause. (Estimated as approximately 1 year)
  Dose Optimization and Safety Lead-In Part B: Number of Participants with a TEAE
Part A and Part B: Progression-Free Survival (PFS) | Randomization to first documented progression of disease or death from any cause. (Estimated as approximately 1 year)
  PFS per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by blinded independent central review (BICR)

SECONDARY OUTCOMES:
Part A and Part B: Overall Survival (OS) | Randomization to date of death from any cause. (Estimated as up to 3 years)
  Part A and Part B: OS
Part A and Part B: PFS | Randomization to first documented progression of disease or death from any cause. (Estimated as approximately 1 year)
  PFS per RECIST v1.1 by investigator
Part A and Part B: Overall Response Rate (ORR): Percentage of Participants who Achieve a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) | Randomization to disease progression or death. (Estimated as approximately 1 year)
  ORR per RECIST v1.1 by BICR and Investigator
Part A and Part B: Duration of Response (DOR) | Date of first evidence of CR or PR to date of disease progression or death from any cause. (Estimated as approximately 1 year)
  DOR per RECIST v1.1 by BICR and Investigator
Part A and Part B: Disease Control Rate (DCR): Percentage of Participants who Achieve a BOR of CR, PR, or Stable Disease (SD) | Randomization to disease progression or death from any cause. (Estimated as approximately 1 year)
  DCR per RECIST v1.1 by BICR and Investigator
Part A and Part B: Time to Response (TTR) | Time from randomization until the date that measurement criteria for CR or PR (whichever is first recorded) are first met (Estimated as approximately 1 year)
  TTR per RECIST v1.1 by BICR and Investigator
Part A and Part B: Intracranial Overall Response Rate (ORR) | Randomization to intracranial disease progression or death. (Estimated as approximately 1 year)
  Intracranial ORR per Modified RECIST (mRECIST) by BICR
Part A and Part B: Intracranial Duration of Response (DoR) | Date of first evidence of CR or PR to date of intracranial disease progression or death from any cause. (Estimated as approximately 1 year)
  Intracranial DoR per mRECIST by BICR
Part A and Part B: PFS2 | Randomization to disease progression on next line of treatment or death from any cause (Estimated as approximately 1 year
  Part A and Part B: PFS2 by Investigator
Part A and Part B: Changes in NSCLC-related symptoms as measured by NSCLC-SAQ | Randomization through end of treatment (Estimated as approximately 1 year)]
  NSCLC-related symptoms are assessed by the NSCLC-SAQ total score, which is computed as the sum of the 5 domains (7 questions) and ranges from 0 to 20. The total score will be calculated if all 7 questions are completed. Higher scores indicate more severe symptomatology.
Part A and Part B: Time to Worsening of NSCLC-related Symptoms as Measured by NSCLC Symptom Assessment Questionnaire (NSCLC-SAQ) | Randomization through end of treatment (Estimated as approximately 1 year)
  NSCLC symptoms will be assessed using the 7-item NSCLC-SAQ. The NSCLC-SAQ measures overall symptom severity of NSCLC, including cough, pain, dyspnea, fatigue, and poor appetite. Response options range from 0) "Not at all" to 4) "Always" or from 0) "Never" to 4) "Always." The total score ranges from 0-20. Higher scores represent worse symptoms.
Part A and Part B: Changes in physical function, as measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (EORTC QLQ-C30) Physical Functioning subscale and IL19 | Randomization through end of treatment (Estimated as approximately 1 year)
  Physical function is assessed by EORTC-QLQ-C30 Physical Functioning scale or IL19. The physical function score is calculated by generating the raw score: (Q1+Q2+Q3+Q4+Q5)/5; and then generating the transformed score: (1-((raw score-1)/3)) x 100. The score ranges from 0 to 100. Higher scores indicate better physical function.
Part A and Part B: Time to Deterioration in Physical Function, as Measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (EORTC QLQ-C30) Physical Functioning Subscale and IL19 | Randomization through end of treatment (Estimated as approximately 1 year)
  The EORTC QLQ-C30 is a 30-question patient-reported instrument used to assess multidimensional health-related quality of life (HRQoL) in cancer patients. Physical functioning is measured by the EORTC-QLQ-30 Physical Function Scale (five items). Response options range from 1) "Not at all" to 4) "Very much." The sum score is linearly transformed to the range 0 - 100. Higher scores represent better physical function.
Part A and Part B: Proportion of Time with High Side-Effect Burden, as Measured by Functional Assessment of Cancer Therapy - General Item 5 (FACT-GP5) | Randomization through end of treatment (Estimated as approximately 1 year)
  FACT-GP5 is a single-item, patient-reported instrument for assessing overall treatment side-effect burden. Response options range from 0) "Not at all" to 4) "Very much." Higher scores represent higher symptom burden.
Part A and Part B: Change from Baseline in Overall Health-related Quality of Life, as Measured by the EORTC QLQ-C30 Global Health Status/Quality of Life Subscale | Randomization through end of treatment (Estimated as approximately 1 year)
  The EORTC QLQ-C30 is a 30-question patient-reported instrument used to assess multidimensional HRQoL in cancer patients. Overall HRQoL is measured by the EORTC QLQ-30 Global Health Status/Quality of Life Subscale (two items). Response options range from 1) "very poor" to 7) "excellent." Scores are linearly transformed to the range 0 - 100. Higher scores represent better overall HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (424):
- United States (91):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mercy Cancer Center, Merced, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - BASS Cancer Center, Walnut Creek, California
  - USO - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Millennium Oncology Research Clinic, Hollywood, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Ocala Oncology Center PL DBA Florida Cancer Affiliates - Ocala, Ocala, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Emory University School of Medicine- Grady Campus, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Hospital, Chicago, Illinois
  - Springfield Clinic Main Campus, Springfield, Illinois
  - Parkview Research Center at Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - The University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - CHI Saint Joseph Cancer Center - East, Lexington, Kentucky
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - USO - Maryland Oncology Hematology, Annapolis, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - The Cancer & Hematology Centers, Grand Rapids, Michigan
  - Allina Health Cancer Institute - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - HealthPartners Cancer Research Center, Saint Paul, Minnesota
  - North Mississippi Hematology and Oncology Associates, Tupelo, Mississippi
  - Oncology Hematology Associates, Springfield, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The Valley Hospital, Inc., Paramus, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Maimonides Cancer Center, Brooklyn, New York
  - Northwell Health/ RJ Zuckerberg Cancer Center, Lake Success, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Manhattan Eye, Ear and Throat Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Clinical Research Alliance, Westbury, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - UNC REX Cancer Center, Raleigh, North Carolina
  - USO - Oncology Hematology Care, Cincinnati, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer -T, Columbus, Ohio
  - USO - Oncology Associates of Oregon, Eugene, Oregon
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Interstate Medical Office Central, Portland, Oregon
  - USO - Alliance Cancer Specialists, PC, Horsham, Pennsylvania
  - Thomas Jefferson University, Sidney Kimmel Cancer Center - Clinical Trials Office, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Lifespan Cancer Institute, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Memorial Hospital-Memphis, Memphis, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - USO - US Oncology Research Network, Nashville, Tennessee
  - USO - Texas Oncology, Austin, Texas
  - William Beaumont Army Medical Center, Fort Bliss, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - USO - Texas Oncology, Webster, Texas
  - The University of Vermont Medical Center Inc., Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - USO - Virginia Cancer Specialists, Fairfax, Virginia
  - VCU Health Adult Outpatient Pavillion, Richmond, Virginia
  - Swedish Cancer Institute - Edmonds, Edmonds, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Swedish Medical Center, Seattle, Washington
  - VA Puget Sound Health Care System, Seattle, Washington
  - USO - Northwest Cancer Specialists, Vancouver, Washington
  - SSM Health Dean Medical Group - South Madison Campus Health Research/Circuit Clinical, Madison, Wisconsin
- Australia (11):
  - Royal Adelaide Hospital, Adelaide
  - Icon Cancer Centre Wesley, Auchenflower
  - Ballarat Health Services, Ballarat Central
  - Sunshine Coast University Hospital, Birtinya
  - Gosford Hospital, Gosford
  - Mackay Base Hospital, Mackay
  - St Vincent's Hospital, Melbourne
  - Sir Charles Gairdner Hospital, Perth
  - Goulburn Valley Health, Shepparton
  - Gold Coast University Hospital, Southport
  - The Townsville Hospital, Townsville
- Austria (3):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Klinik Floridsdorf, Vienna
- Belgium (10):
  - ZNA Middelheim, Antwerp
  - CHIREC - site delta, Auderghem
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - UZ Gent, Ghent
  - AZ Groeninge Campus Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - AZ Sint-Maarten, Mechelen
  - Clinique Saint Pierre, Ottignies
  - AZ Glorieux Ronse, Ronse
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godinne, Yvoir
- Brazil (29):
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos
  - Hospital Tacchini, Bento Gonçalves
  - Hospital São Domingos, Bequimão
  - Sirio-Libanes Brasilia - Centro de Oncologia - Asa Sul, Brasília
  - Hospital Universitário Evangélico Mackenzie, Curitiba
  - Centro de Pesquisa Clínica do Instituto do Câncer do Ceará, Fortaleza
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí
  - Hospital Brasilia, Lago Sul
  - Hospital de Cancer de Londrina, Londrina
  - Liga Norte Riograndense Contra o Câncer, Natal
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Oncominas, Pouso Alegre
  - Instituto Nacional de Câncer José Alencar Gomes da Silva - INCA, Rio de Janeiro
  - Centro de Tratamento de Tumores Botafogo para Oncoclinicas Rio de Janeiro SA, Rio de Janeiro
  - Instituto D'Or Pesquisa e Ensino, Rio de Janeiro
  - Clinica Amo - Rio Vermelho, Salvador
  - Faculdade de Medicina do ABC, Santo André
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - COE Ensino e Pesquisa, São José dos Campos
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
  - Hospital Sírio Libanês, São Paulo
  - Hospital Santa Catarina - Paulista, São Paulo
  - Hospital BP, São Paulo
  - Hospital Paulistano, São Paulo
  - Centro Paulista de Oncologia Clínica, São Paulo
  - Núcleo de Pesquisa Clínica da Rede São Camilo, São Paulo
  - Instituto de Assistência Médica ao Servidor Público Estadual - IAMSPE/HSPE-FMO Conhecer Centro de Oncolog -T, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo
  - CEDOES, Vitória
- Canada (3):
  - BC Cancer Abbotsford, Abbotsford
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi
  - BC Cancer Vancouver, Vancouver
- China (35):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing
  - Beijing Cancer hospital, Beijing
  - Jilin Province Tumor Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - The First People's Hospital of Changzhou, Changzhou
  - The Third People's Hospital of Chengdu (CDTPH), Chengdu
  - Sichuan Cancer hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Hainan General Hospital, Haikou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jinan Central Hospital, Jinan
  - Shandong Cancer Hospital, Jinan
  - Taizhou Hospital of Zhejiang Province, Linhai
  - LinYi Cancer Hospital, Linyi
  - Liuzhou People's Hospital, Liuchow
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing First Hospital, Nanjing
  - Nantong Tumor Hospital, Nantong
  - Shanghai Chest Hospital, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Xinjiang Medical University Cancer Hospital - Urumqi, Ürümqi
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan
  - Wuhan Union Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wannan Medical College Yijishan Hospital, Wuhu
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xiangyang Central Hospital, Xiangyang
  - Yichang Central People's Hospital, Yichang
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang
  - ZhuZhou Central Hospital, Zhuzhou
- Czechia (2):
  - Nemocnice AGEL Ostrava - Vitkovice a.s., Ostrava
  - Fakultni nemocnice Bulovka, Prague
- Roskilde University Hospital, Roskilde, Denmark
- France (18):
  - Sainte Catherine Institut du Cancer Avignon Provence, Avignon
  - Hospices Civils de Lyon - Hopital Louis Pradel, Bron
  - CHU Lille - Institut Coeur Poumon, Lille
  - Centre Leon Berard, Lyon Cedex08
  - Centre Antoine-Lacassagne, Nice
  - Institut Curie, Paris
  - CHU Bordeaux Haut-Leveque, Pessac
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Nouvel Hôpital Civil (NHC), Strasbourg
  - Hôpital Foch, Suresnes
  - Centre Hospitalier intercommunal de Toulon La Seyne sur Mer, Toulon
  - CHU de Toulouse - Hopital Larrey, Toulouse
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - Hôpital Robert Schuman, Vantoux
  - Gustave Roussy, Villejuif
- Germany (18):
  - Evangelische Lungenklinik Berlin, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Helios Klinikum Emil von Behring Berlin-Zehlendorf, Berlin
  - Klinikum Chemnitz, Chemnitz
  - MV-Zentrum für Onkologie und Hämatologie, Cologne
  - Onkologiezentrum Donauwörth, Donauwörth
  - HELIOS Klinikum Erfurt, Erfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Fachkliniken München-Gauting, Gauting
  - Franziskus-Hospital Harderberg, Georgsmarienhütte
  - LungenClinic Grosshansdorf, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Dölau, Halle
  - Hämato-Onkologie Hamburg, Prof. Laack und Partner, Hamburg
  - Asklepios Klinik Harburg, Hamburg
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster
  - Klinikum Nürnberg Nord, Nuremberg
  - Universitaetsklinikum Tuebingen, Tübingen
- Greece (9):
  - Agios Savvas Regional Cancer Hospital, Athens
  - Errikos Dunant Hospital Center, Athens
  - Sotiria Thoracic Diseases Hospital of Athens, Athens
  - Attikon General University Hospital, Chaïdári
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Patras, Pátrai
  - "Theagenio" Cancer Hospital of Thessaloniki, Thessaloniki
  - European Interbalkan Medical Center, Thessaloniki
  - G. Papanikolaou General Hospital, Thessaloniki
- Hungary (5):
  - Országos Korányi Pulmonológiai Intézet, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
  - Farkasgyepui Tudogyogyintezet, Farkasgyepű
  - Bacs-Kiskun Megyei Korhaz, Kecskemét
- India (18):
  - Hemato Oncology Clinic, Ahmedabad
  - KLES Dr. Prabhakar Kore Hospital & M.R.C, Belagavi
  - SRV Hospitals, Bengaluru
  - All India Institute of Medical Sciences, Bhubaneswar
  - Ashwin Hospital, Coimbatore
  - Nizam's Institute of Medical Sciences, Hyderabad
  - Krishna Institute of Medical Sciences - Karad, Karad
  - Kolhapur Cancer Centre Private Limited, Kolhāpur
  - Tata Memorial Hospital, Mumbai
  - HCG Manavata Cancer Centre, Nashik
  - Jawaharlal Institute Of Postgraduate Medical Education And Research, Puducherry
  - Grant Medical Foundation - Ruby Hall Clinic, Pune
  - Sahyadri Super Speciality Hospital, Pune
  - Lifepoint Multispeciality Hospital, Pune
  - Regional Cancer Centre - Thiruvananthapuram, Thiruvananthapuram
  - Pacific Medical College & Hospital, Udaipur
  - Tata Memorial Centre - Homi Bhabha Cancer Hospital, Varanasi
  - Mahatma Gandhi Cancer Hospital and Research Institute, Visakhapatnam
- Italy (10):
  - Instituto Tumori Giovanni Paolo II, Bari
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Policlinico "G. Rodolico", Catania
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Istituto Nazionale Tumori Regina Elena, Rome
  - Ospedale di Circolo e Fondazione Macchi Varese, Varese
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona
- Japan (30):
  - National Hospital Organization Asahikawa Medical Center, Asahikawa
  - Juntendo University Hospital, Bunkyō City
  - Tokyo Metropolitan Komagome Hospital, Bunkyō City
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka
  - Himeji Medical Center, Himeji
  - Kansai Medical University Hospital, Hirakata
  - Kanazawa University Hospital, Kanazawa
  - Ibaraki Prefectural Central Hospital, Kasama
  - National Cancer Center Hospital East, Kashiwa
  - Kobe City Medical Center General Hospital, Kobe
  - Japanese Foundation for Cancer Research, Kōtō City
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Shizuoka Cancer Center, Nagaizumi-cho,Sunto-gun
  - Nagasaki University Hospital, Nagasaki
  - Aichi Cancer Center Hospital, Nagoya
  - Miyagi Cancer Center, Natori
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Kindai University Hospital- Osakasayama Campus, Sakai
  - National Hospital Organization Kinki-chuo Chest Medical Center, Sakai
  - Hokkaido University Hospital, Sapporo
  - National Hospital Organization Yamaguchi Ube Medical Center, Ube
  - Tochigi Cancer Center, Utsunomiya
  - Wakayama Medical University Hospital, Wakayama
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
  - Kanagawa cancer center, Yokohama
  - Tottori University Hospital, Yonago
- Mexico (15):
  - CIO - Centro de Inmuno-Oncología de Occidente, Guadalajara
  - PanAmerican Clinical Research - Guadalajara, Guadalajara
  - Actualidad Basada en la Investigación del Cáncer, Guadalajara
  - Renati Innovation, Guadalajara
  - Health Pharma Querétaro, Juriquilla
  - Preparaciones Oncológicas S.C., León
  - Health Pharma Professional Research S.A. de C.V:, Mexico City
  - Centro Onco-Hematológico Roma (COHR), Mexico City
  - Higiea Oncologia, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey
  - Avix Investigación Clinica, S.C., Monterrey
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
  - Clinica Integral Internacional de Oncología, Puebla City
  - Oncare - Unidad Valle, San Pedro Garza García
  - Arké SMO S.A de C.V, Veracruz
- Netherlands (9):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Medisch Spectrum Twente, Enschede
  - Ziekenhuis St. Jansdal, Harderwijk
  - Tergooiziekenhuizen, locatie Hilversum, Hilversum
  - Frisius Medisch Centrum, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus Medisch Centrum, Rotterdam
  - ETZ Elisabeth, Tilburg
  - St. Antonius Ziekenhuis, locatie Utrecht, Utrecht
- Norway (7):
  - Haukeland Universitetssjukehus, Bergen
  - Drammen Sykehus, Vestre Viken HF, Drammen
  - Sykehuset Innlandet HF Gjøvik, Gjøvik
  - Akershus Universitetssykehus, Lørenskog
  - Oslo universitetssykehus, Radiumhospitalet, Oslo
  - Stavanger Universitetssykehus, Stavanger
  - St. Olavs Hospital, Trondheim
- Poland (3):
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Kielce
  - One Day Med, Szczecin
  - MICS Centrum Medyczne Torun, Torun
- Portugal (7):
  - Centro Hospitalar E Universitário De Coimbra, Coimbra
  - Champalimaud Foundation, Lisbon
  - Hospital da Luz Lisboa, Lisbon
  - Hospital Pulido Valente, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
  - Hospital CUF Porto, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (8):
  - Lotus-Med, Bucharest
  - SC Memorial Healthcare International SRL, Bucharest
  - Gral Medical Diagnostic Center, Bucharest
  - Institutul Oncologic, Cluj-Napoca
  - Centrul de Oncologie "Sfântul Nectarie", Craiova
  - Ovidius Clinical Hospital OCH, Ovidiu
  - S C Oncocenter Oncologie Clinica S R L, Timișoara
  - Cabinet Medical Oncomed, Timișoara
- South Korea (15):
  - Chungbuk National University Hospital, Cheongju-si
  - Keimyung University Dongsan Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Deagu
  - Gangnam Severance Hospital, Yonsei University Health System, Gangnam-gu
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Hwasun
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University Of Korea St. Vincent's Hospital, Suwon
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (20):
  - CHUAC-Hospital Teresa Herrera, A Coruña
  - Hospital Infanta Cristina, Badajoz
  - OSI Ezkerraldea-Enkarterri-Cruces - Hospital Universitario Cruces, Barakaldo
  - Parc de Salut Mar - Hospital del Mar, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, Hospitalet
  - Hospital Jerez de la Frontera, Jerez de la Frontera
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Complejo Asistencial Universitario de León - Hospital de León, León
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - H.R.U Málaga - Hospital General, Málaga
  - Hospital Universitari Son Espases, Palma
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico de Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- Sweden (2):
  - Mälarsjukhuset, Eskilstuna
  - Västmanlands Sjukhus Västerås, Västerås
- Switzerland (3):
  - CHUV (centre hospitalier universitaire vaudois), Lausanne
  - Kantonsspital Winterthur, Winterthur
  - UniversitätsSpital Zürich, Zurich
- Taiwan (17):
  - Changhua Christian Hospital, Changhua County
  - Buddhist Dalin Tzu Chi General Hospital, Chiayi City
  - National Taiwan University Hospital Yun-Lin Branch Dou-Liou Region, Douliu
  - Hualien Tzu Chi Medical Center, Hualien City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - New Taipei Municipal TuCheng Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - Chi Mei Hospital - Liouying Branch, Tainan
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Cancer Center (NTUCC), Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
  - National Taiwan University Hospital - Hsinchu branch, Zhubei
- Turkey (Türkiye) (17):
  - Adana Medical Park Seyhan Hastanesi, Adana
  - Adana City Hospital, Adana
  - Ankara Etlik City Hospital, Ankara
  - Abdurrahman Yurtaslan Ankara Oncology, education and Research Hospital, Ankara
  - Ankara Bilkent Şehir Hastanesi, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Memorial Antalya Hospital, Antalya
  - Antalya Egitim ve Arastırma Hastanesi, Antalya
  - Uludag Universitesi, Bursa
  - Dicle Üniversitesi, Diyarbakır
  - Bezmialem Vakf Üniversitesi, Istanbul
  - İ.A.Ü VM Medical Park Florya Hastanesi, Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Ege Universitesi Hastanesi, Izmir
  - zmir Katip Çelebi Üniversitesi Atatürk Eitim Ve Aratrma Hastanesi, Izmir
  - Kocaeli Üniversitesi, Kocaeli
  - Ondokuz Mayıs Universitesi, Samsun
- United Kingdom (8):
  - Aberdeen Royal Infirmary, Aberdeen
  - Ninewells Hospital and Medical School, Dundee
  - Huddersfield Royal Infirmary, Huddersfield
  - St James's University Hospital, Leeds
  - The Christie NHS Foundation Trust, Manchester
  - Mount Vernon Hospital, Northwood
  - Weston Park Hospital, Sheffield
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY3537982 Plus Immunotherapy With or Without Chemotherapy in Participants With Non-Small Cell Lung Cancer (NSCLC) With a Change in a Gene Called KRAS G12C (SUNRAY-01) — https://trials.lilly.com/en-US/trial/433515